CLINICAL TRIAL: NCT02720393
Title: Impact of no Carrageenan Diet on Glucose Tolerance in Prediabetes
Brief Title: Impact of No-carrageenan Diet on Glucose Tolerance in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Joanne Kramer Tobacman, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015-1255
Record Dates: First submitted 2016-02-09; First posted 2016-03-25 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular diet (Placebo Comparator): Meals and snacks will contain carrageenan in the amount consumed in the typical daily diet and will be selected by the study dietician and distributed to study subjects randomized to the regular diet study arm.
  Interventions: Other: Regular Diet
- No-carrageenan diet (Experimental): No-carrageenan diet will be composed of meals and snacks selected by the study dietician and distributed to study participants who are randomized to the no-carrageenan diet study arm.
  Interventions: Other: No-carrageenan diet

INTERVENTIONS:
Other: No-carrageenan diet — Diet of food items that have no carrageenan as selected by study dietician.
  Arms: No-carrageenan diet
Other: Regular Diet — Diet of food items that have carrageenan as selected by study dietician
  Other Names: Carrageenan-containing diet
  Arms: Regular diet

SUMMARY:
Participants will be randomly assigned to either regular or no-carrageenan prepared diets to determine whether the no-carrageenan leads to improvement in glucose tolerance. Hemoglobin A1c is the primary outcome measure.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to a diet. They will at onset have hemoglobin A1c values between 5.7% and 6.4%. Baseline glucose tolerance test will be performed, as well as measures of inflammation and fecal microbiome. Interim tests will be performed at six weeks. Subjects will participate for 12 weeks, at which time they will be re-evaluated.

ELIGIBILITY:
Inclusion Criteria:

* per diabetes, ability to follow diet and study procedures

Exclusion Criteria:

* on any medications that affect glucose, medical conditions or allergies that affect adherence to study diet, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c | baseline, 12 weeks
  Measurements performed after 12 weeks of dietary intervention

SECONDARY OUTCOMES:
Change in serum Interleukin-8 | baseline, 12 weeks
  Impact of diet on serum Interleukin-8
Impact on glucose tolerance test | 12 weeks
  perform repeat oral glucose tolerance test after 12 weeks of dietary intervention
Impact on insulin level | 12 weeks
  determine effect of dietary intervention on insulin level at the time of glucose tolerance test
Change in leukocyte subsets | baseline, 12 weeks
  determine if there is change in distribution of leukocyte subsets from blood samples of study participants
Change in Tumor Necrosis Factor-alpha in serum | baseline, 12 weeks
  determine if there is change in circulating TNF-alpha in blood samples
Change in insulin signaling pathway | baseline, 12 weeks
  determine if there are changes in activation of intermediates in insulin signaling pathway in circulating leukocytes following dietary intervention

OTHER OUTCOMES:
Change in fecal microbiome | baseline, 12 weeks
  Impact of diet on fecal microbiome following dietary intervention determined by whole genome sequencing of fecal bacteria
Change in fecal calprotectin | baseline, 12 weeks
  determine effect of dietary intervention on fecal calprotectin

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
If required, individual data without identifiers may be made available.